CLINICAL TRIAL: NCT00316342
Title: Workplace Based Rehabilitation for Low Back Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: The UAW-GM National Joint Committee on Health & Safety (Unknown)
Responsible Party: Dr. Gunnar Andersson, Rush University Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 95050341; #97-1-AP
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain
Keywords: Low back pain; Industrial workers; Recurrent back pain; Back supports; Back health education; Rehabilitation
MeSH Terms: conditions — Low Back Pain; Back Pain

INTERVENTIONS:
Device: Back supports

SUMMARY:
The purpose of this study is to examine the effect of back supports plus education upon recovery from a work-related low back disorder. The study tests the hypothesis: the use of back supports plus health education is not different from health education alone in promoting recovery from a work-related low back disorder in consideration of personal, health, and job factors. Significant improvements in physical health, neurogenic symptoms, back pain disability, and low back pain were observed over the twelve months of study follow-up. No statistically significant difference between the study groups was found with respect to these measures.

DETAILED DESCRIPTION:
BACKGROUND Low back pain remains a common major source of morbidity and disability. Few studies consider the effectiveness of interventions for low back pain while simultaneously considering personal, health, and job characteristics.

METHODS This is a randomized clinical trial in which 433 active employees with low back disorders were randomly assigned to one of two study groups: 1) back support plus education on back health; or 2) education on back health only. Demographic, health, medical, and job factors were recorded. Outcomes were evaluated over a twelve month period and included self-reported measures of back pain, back pain disability level, physical health, mental health, back pain recurrence and administrative measures.

RESULTS Significant improvements in physical health, neurogenic symptoms, back pain disability, and low back pain were observed over time in both study groups. However, there was no significant difference between the study groups with respect to these outcome measures. The adjusted hazard ratio of recurrence rate was suggestive of an incremental protective effect due to back supports over education alone (adjusted hazard ratio [AHR]=0.711, 95% CI 0.50, 1.04, p=.085). There was also a marginal effect of back supports and education on decreasing low back pain over time (AHR=0.0015, p=0.091).

CONCLUSIONS Back supports may have some value in promoting recovery from low back pain, but this effect is only observed in individuals who are actively employed in jobs with medium risk of low back disorders.

ELIGIBILITY:
Inclusion Criteria:

work-related low back disorder, 18-64 years of age,active hourly worker, enrollment into study within eight weeks of diagnosis, signed informed consent

Exclusion Criteria:

no other concurrent work-related condition not pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 433
Dates: Start 1997-01; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Low back pain
Back pain disability
Neurogenic symptoms
Physical health
Mental health
Low back pain repeated episodes
Lost work time

CONTACTS AND LOCATIONS:
Overall Officials: Denise M Oleske, PhD, Principal Investigator — Rush University Medical Center

REFERENCES:
- [Background] Oleske DM, Lavender SA, Andersson GB, Morrissey MJ, Zold-Kilbourn P, Allen C, Taylor E. Risk factors for recurrent episodes of work-related low back disorders in an industrial population. Spine (Phila Pa 1976). 2006 Apr 1;31(7):789-98. doi: 10.1097/01.brs.0000207017.30490.28. PMID 16582853
- [Background] Oleske DM, Neelakantan J, Andersson GB, Hinrichs BG, Lavender SA, Morrissey MJ, Zold-Kilbourn P, Taylor E. Factors affecting recovery from work-related, low back disorders in autoworkers. Arch Phys Med Rehabil. 2004 Aug;85(8):1362-4. doi: 10.1016/j.apmr.2003.11.021. PMID 15295767
- [Background] Oleske D, Lavender S, Andersson G, Hahn J, Zold-Kilbourn P, Allen-Toole C, Laskowski J. Job exposures as correlates of recovery in population-based rehabilitation intervention for work-related low back disorders. Ann Epidemiol. 2000 Oct 1;10(7):481. doi: 10.1016/s1047-2797(00)00165-4. PMID 11018430
- [Background] Oleske DM, Andersson GB, Lavender SA, Hahn JJ. Association between recovery outcomes for work-related low back disorders and personal, family, and work factors. Spine (Phila Pa 1976). 2000 May 15;25(10):1259-65. doi: 10.1097/00007632-200005150-00010. PMID 10806503
- [Background] Lavender SA, Oleske DM, Nicholson L, Andersson GB, Hahn J. Comparison of five methods used to determine low back disorder risk in a manufacturing environment. Spine (Phila Pa 1976). 1999 Jul 15;24(14):1441-8. doi: 10.1097/00007632-199907150-00009. PMID 10423789